CLINICAL TRIAL: NCT04715880
Title: The Comparison of the Analgesic Efficacy and Hemodynamic Effects of Paravertebral Block Compared With Paravertebral and Intercostal Nerve Block for Thoracotomy in Adults: A Randomized Controlled Trail
Brief Title: The Comparison of the Analgesic Efficacy and Hemodynamic Effects of Paravertebral Block Compared With Paravertebral and Intercostal Nerve Block for Thoracotomy in Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Kumar Sundeep, Trainee Medical Officer Anaesthesiology, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-0797-7328
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Pain, Postoperative; Nerve Block; Thoracotomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Population Groups; PVB protocol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral Block (PVB) group (Active Comparator): Under complete aseptic precaution, Patient will be in lateral decubitus position a paravertebral catheter will be placed by the surgeon before closure of thoracotomy wound. The catheter will be introduced percutaneously through 18 gauge needle into the pleural cavity.
  The tip of catheter will be loaded by anaesthesiologist with 0.25 % isobaric bupivacaine with 20 ml followed by continuous infusion with bupivacaine 0.25 % at 6-8 ml per hour
  Interventions: Procedure: Paravertebral Block (PVB) group
- Paravertebral block/Intercostal Block (PVB/ICB) group (Active Comparator): Under complete aseptic precaution, patient will be in lateral decubitus position a paravertebral catheter will be placed by surgeon into pleural cavity and will not be loaded with bolus dose. At the end of surgery the (consultant anaesthesiologist) will perform intrathoracic unilateral intercostal nerve block two level above and two level below and at site of incision with 4 ml per level of 0.25 % bupivacaine followed by continuous infusion with 0.25 % bupivacaine at 6-8 ml/hour through catheter placed in paravertebral space.
  Interventions: Procedure: Paravertebral block/Intercostal Block (PVB/ICB) group

INTERVENTIONS:
Procedure: Paravertebral block/Intercostal Block (PVB/ICB) group — A paravertebral catheter will be placed by surgeon into pleural cavity and will not be loaded with bolus dose. At the end of surgery the (consultant anaesthesiologist) will perform intrathoracic unilateral intercostal nerve block two level above and two level below and at site of incision with 4 ml per level of 0.25 % bupivacaine followed by continuous infusion with 0.25 % bupivacaine at 6-8 ml/hour through catheter placed in paravertebral space.
  Arms: Paravertebral block/Intercostal Block (PVB/ICB) group
Procedure: Paravertebral Block (PVB) group — A paravertebral catheter will be placed by the surgeon before closure of thoracotomy wound. The catheter will be introduced percutaneously through 18 gauge needle into the pleural cavity. The tip of catheter will be loaded by anaesthesiologist with 0.25 % isobaric bupivacaine with 20 ml followed by continuous infusion with bupivacaine 0.25 % at 6-8 ml per hour
  Arms: Paravertebral Block (PVB) group

SUMMARY:
Thoracotomy is a surgical procedure associated with severe post operative pain during the first day of surgery and is responsible for prolonged hospital stay, patient dissatisfaction and delayed return to normal activities along with increased morbidity and mortality. Investigators intend to compare the efficacy of two analgesic interventions (continuous infusion of paravertebral block (PVB) after loading dose compared with intercostal nerve block and continuous infusion of PVB without loading dose) on postoperative thoracotomy pain. The results of this study will direct the investigators to find the best practice methods which will reduce the postoperative thoracotomy pain, the overall cost of pain management and length of patient's hospital stay.

DETAILED DESCRIPTION:
Objective To compare the safety, efficacy for pain relief and hemodynamic changes of two analgesic interventions(continuous infusion of Paravertebral block (PVB) after loading dose compared with intercostal nerve block and continuous infusion of PVB without loading dose)

ELIGIBILITY:
Inclusion Criteria:

* All ASA I-IV adult patients between the ages of 18-70 years scheduled for elective thoracotomy
* Either sex

Exclusion Criteria:

1. Neurological or psychiatric diseases
2. Emergency Procedures.
3. Language barrier
4. Patients under chronic treatment with opioids
5. Patients with hypersensitivity to bupivacaine
6. Coagulation disorders.
7. Unwilling to participate.
8. Patient previously involved in other studies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Pain Score | 24 hours
  Visual Analogue Scale (VAS) pain Score in cm (0cm = No pain and 10 cm= Worst pain possible)
Blood Pressure | 24 hours
  Blood pressure in mmHg
Heart Rate | 24 Hours
  Heart rate per minute

SECONDARY OUTCOMES:
Total postoperative narcotic consumption | 24 hours
  Patient controlled intravenous analgesia (PCIA) nalbuphine or Tramadol consumption in mg
Sedation score | 24 hours
  Ramsay sedation scale: 1= anxious or restless, or both, 2 = Co-operative, oriented, and tranquil, 3 = Responding to commands, 4 = brisk response to stimulus, 5 = sluggish response to stimulus, 6 = no response to stimulus

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perttunen K, Nilsson E, Heinonen J, Hirvisalo EL, Salo JA, Kalso E. Extradural, paravertebral and intercostal nerve blocks for post-thoracotomy pain. Br J Anaesth. 1995 Nov;75(5):541-7. doi: 10.1093/bja/75.5.541. PMID 7577277
- [Background] Yeung JH, Gates S, Naidu BV, Wilson MJ, Gao Smith F. Paravertebral block versus thoracic epidural for patients undergoing thoracotomy. Cochrane Database Syst Rev. 2016 Feb 21;2(2):CD009121. doi: 10.1002/14651858.CD009121.pub2. PMID 26897642
- [Derived] Kumar S, Hameed M, Shehzad R, Samad K. The comparison of the analgesic efficacy of continuous paravertebral block alone compared with continuous paravertebral and intercostal nerve block for thoracotomy in adults: a randomized controlled trial. J Anesth. 2023 Dec;37(6):923-929. doi: 10.1007/s00540-023-03255-8. Epub 2023 Sep 25. PMID 37747499